CLINICAL TRIAL: NCT03207594
Title: Improving Evidence-Based Care for Cancer Patients
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 102472
Record Dates: First submitted 2017-03-22; First posted 2017-07-05 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Cancer; Prostate Cancer; Breast Cancer; Lung Cancer; Gynecologic Cancer; Gastrointestinal Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Prostatic Neoplasms; Breast Neoplasms; Lung Neoplasms; Gastrointestinal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Arm 1: Current smokers with cancer who are planning to get radiation therapy at MUSC.
  Interventions: Other: Survey; Other: Saliva sample; Other: Smoking Status questions

INTERVENTIONS:
Other: Survey — Subjects will be asked to complete a survey asking questions about his/her current health, well-being and quality of life.
Other: Saliva sample — Subjects will have saliva collected by a member of the study team using a cotton swab.
Other: Smoking Status questions — Subjects will be asked to complete an assessment asking questions about his/her current smoking status

SUMMARY:
The purpose of this study is to improve cancer care and the delivery of cancer care. Researchers are interested in studying patient reported information and examining how different factors may impact cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with head/neck, lung, breast, prostate, gastrointestinal or gynecologic cancer
* 21 years of age or older at time of study registration
* Must have been referred to MUSC radiation oncology for treatment with curative radiation therapy
* Must report current smoking defined as self-reporting smoking within the past 30 days using a structured intake questionnaire.

Exclusion Criteria:

* Patients with primary central nervous system malignancies will be excluded.
* Patients that have other cancer disease types will be excluded due to either significant differences in standard radiation therapy approaches or rarity of disease required radiation.
* Patients who are currently participating in the Medical University of South Carolina Hollings Cancer Center smoking cessation program
* Patients who are unable to provide informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who have been diagnosed with head/neck, lung, breast, prostate, gastrointestinal or gynecologic cancers that are 21 years of age or older. Patients must have been referred to MUSC radiation oncology for treatment with curative radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with biochemically confirmed smoking cessation | 4 weeks after enrollment
  Biochemical confirmation will be determined by saliva samples
Number of patient who self-report smoking cessation | 4 weeks after enrollment
  Self-reported smoking cessation will be documented via smoking assessment questionnaire

SECONDARY OUTCOMES:
Average weekly smoke exposure | up to 62 weeks
  reported cigarettes per day multiplied by the number of days smoked during radiation therapy (RT), summed over a period of time and normalized to yield an average weekly smoke exposure during RT.
Number of patients who participate in smoking cessation | up to 12 months after completion of RT.
  Completing one in-person visit where an individualized smoking cessation treatment plan is developed and implemented.
Compliance with smoking cessation | up to 12 weeks after completion of RT
  Two binary measure of compliance:
  1. - completing at least three in person visits within 6 weeks of starting an individualized cessation treatment plan
  2. - completing at least one in-person visit and at least two phone-based communications

CONTACTS AND LOCATIONS:
Overall Officials: Graham Warren, MD, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No